CLINICAL TRIAL: NCT06412848
Title: A Multicenter, Retrospective, Observational Study of Avelumab Maintenance and Subsequent Therapies in Japanese Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: JAVEMACS: Japan AVElumab Maintenance And Continuous Treatment Study
Status: Active, not recruiting | Type: Observational
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: MS100070_0209
Record Dates: First submitted 2024-04-23; First posted 2024-05-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial Carcinoma; Avelumab; JAVEMACS; Locally advanced UC; Metastatic UC
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — avelumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Urothelial Carcinoma Cohort: This is a single cohort study enrolling Participants with Urothelial Carcinoma (UC), who are prescribed treatment with avelumab as first line maintenance therapy after a platinum-based chemotherapy (PBCT).
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — This is an observational study, participants who received avelumab as first line maintenance therapy after a PBCT.

SUMMARY:
This study is a multicenter, non-interventional, retrospective, medical chart review of locally advanced or metastatic (la/m) Urothelial Cancer UC participants who were prescribed avelumab as first line maintenance therapy after a platinum-based chemotherapy. This study aims to understand the index date (i.e., at the initiation of avelumab maintenance therapy) demographics and clinical characteristics of participants with locally advanced/metastatic Urothelial Carcinoma in Japan, and to describe their treatment patterns and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with locally advanced/metastatic urothelial carcinoma (la/m UC) before receiving avelumab first line maintenance therapy
* Participants with la/m UC (irrespective of tumor histology) whose disease has not progressed (ongoing stable disease, partial response, or complete response) following completion of first line PBCT and who has been treated with avelumab
* Participants who has been started avelumab first line maintenance therapy for la/m UC from 24 Feb 2021 (date of approval for UC) to 6 months before the date of approval of implementation of this study at each site
* Participants aged >= 18 years old at index date
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participant participated in a clinical trial in la/m UC during the study periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with locally advanced/metastatic Urothelial Carcinoma
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Baseline clinical and demographic characteristics | Baseline
  To describe the baseline clinical and demographic characteristics of participants.
Characteristics of the first line PBCT just prior to avelumab maintenance | Up to 3 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 3 months
Progression-Free Survival (PFS) | Up to 3 months
Time to Treatment Failure (TTF) | Up to 3 months
Time to Next Treatment (TTNT) | Up to 3 months
Objective Response Rate (ORR) | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (26):
- Japan (26):
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Ehime University Hospital, Tōon, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Nara Medical University Hospital, Kashihara, Nara
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Juntendo University Hospital, Bunkyō City, Tokya
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Akita University Hospital, Akita
  - Kyushu Cancer Center, Fukuoka
  - Kumamoto University Hospital, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Osaka International Cancer Institute, Osaka
  - Tokushima University Hospital, Tokushima
  - Toyama University Hospital, Toyama
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial Awareness and Transparency Website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100070_0209
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html